CLINICAL TRIAL: NCT07174596
Title: Evaluation of Approved Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6617
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control/Control (Experimental): Eligible subjects will be randomized to the test/control/control sequence, to wear the test lens, the control lens, and the control lens again for 1-week each in a daily disposable modality for at least 5 days per week and 6 hours per day.
  Interventions: Device: B+L Infuse spherical soft contact lenses; Device: J&J ACUVUE OASYS 1-Day spherical soft contact lenses
- Control/Test/Test (Experimental): Eligible subjects will be randomized to the control/test/test sequence, to wear the control lens, the test lens, and the test lens again for 1-week each in a daily disposable modality for at least 5 days per week and 6 hours per day.
  Interventions: Device: B+L Infuse spherical soft contact lenses; Device: J&J ACUVUE OASYS 1-Day spherical soft contact lenses

INTERVENTIONS:
Device: B+L Infuse spherical soft contact lenses — Test lens
Device: J&J ACUVUE OASYS 1-Day spherical soft contact lenses — Control lens

SUMMARY:
This is a prospective, randomized, controlled, subject-masked, bilateral, dispensing, multi-site, 2 lenses × 3 wearing periods crossover study to evaluate visual acuity.

ELIGIBILITY:
Potential subjects must satisfy all of the following criteria to be enrolled in the study: 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.

2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.

3. Be between 18 and 39 (inclusive) years of age at the time of screening. 4. By self-report, habitually wear spherical soft silicone hydrogel contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.

5. Have a habitual contact lens prescription that is current (no power change needed) within the prior 6 months, and they must have worn that prescription for at least 2 weeks prior to entering the study.

6. Possess a wearable pair of spectacles that provide correction for distance vision.

7. The spherical equivalent of the subject's vertex-corrected distance refraction must be between -1.00 D and -6.00 D in each eye.

8. The best corrected, monocular, distance visual acuity must be 20/25 or better in each eye.

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Be currently using any ocular medications or have any ocular infection of any type.
3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See Section 9.1 for additional details regarding excluded systemic medications.
4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
5. Be currently wearing monovision or multifocal contact lenses.
6. Be currently wearing lenses in an extended wear modality.
7. Have a known hypersensitivity or allergic reaction to silicone hydrogel soft contact lenses.
8. Have participated in a contact lens or lens care product clinical trial within 14 days prior to study enrollment.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities, or bulbar injection) or other corneal or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
11. Have a history of strabismus or amblyopia.
12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2025-09-11 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Proportion of Eyes Achieving 20/20 Distance Monocular Snellen VA or Better at the 1-week follow-up visit | At 1-week follow-up per wear period
  Visual acuity (VA) will be collected for each eye at distance using Snellen charts at the fitting evaluation and after approximately 1-week of lens wear.
Proportion of Eyes with acceptable lens fit | Up to 3-week follow-up
  Acceptable lens fit will be assessed at all study visits (scheduled and unscheduled) for each eye.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (4):
- United States (4):
  - VisualEyes, Roswell, Georgia
  - New Bremen EyeCare, New Bremen, Ohio
  - Botetourt Eyecare LLC, Salem, Virginia
  - New River Vision Care, Oak Hill, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu